CLINICAL TRIAL: NCT06498180
Title: A Randomized Self-control Study of Periodontal Initial Treatment Under Local Anesthesia Combined With Glucocorticoid Therapy for Erosive Oral Lichen Planus
Brief Title: Periodontal Initial Treatment Combined With Glucocorticoid Therapy for Erosive Oral Lichen Planus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-T69-OLP-CP
Record Dates: First submitted 2024-07-07; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-04

CONDITIONS: Oral Lichen Planus; Periodontal Diseases
Keywords: Periodontal initial therapy; Erosive oral lichen planus; Local anesthesia
MeSH Terms: conditions — Lichen Planus, Oral; Periodontal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): In the experimental group, subjects will undergo periodontal initial treatment under local anesthesia combined with glucocorticoid local blockade therapy (such as triamcinolone acetonide injection), local use of triamcinolone acetonide ointment, and 1% sodium bicarbonate rinse (avoiding systemic use during visits) after baseline examination, while receiving the following professional oral hygiene guidance:
  Instructions and demonstrations for using manual toothbrushes Instructions and demonstrations for using dental floss or interdental brushes A periodontist with rich clinical experience will perform periodontal initial treatment under local anesthesia.
  Interventions: Other: Periodontal initial treatment under local anesthesia; Drug: Glucocorticoid Therapy; Behavioral: oral hygiene instruction
- Control group (Active Comparator): In the control group, participants will undergo routine glucocorticoid local blockade therapy (such as triamcinolone acetonide injection), local administration of triamcinolone acetonide ointment, and 1% sodium bicarbonate rinse (avoiding systemic medication during visits) after baseline examination, while receiving the following professional oral hygiene guidance:
  Instructions and demonstrations for using manual toothbrushes Instructions and demonstrations for using dental floss or interdental brushes Based on ethical considerations, all participants will receive full mouth periodontal initial treatment at the end of the trial.
  Interventions: Drug: Glucocorticoid Therapy; Behavioral: oral hygiene instruction

INTERVENTIONS:
Other: Periodontal initial treatment under local anesthesia — Removal of plaque retention factors, supragingival scaling and subgingival scraping under local anesthesia with articaine (combined with manual and ultrasound methods), and polishing
  Arms: Experimental group
Drug: Glucocorticoid Therapy — Local blockade therapy with Betamethasone Sodium Phosphate Injection (containing 1.4mg Betamethasone equivalent), local use of 1% Triamcinolone Acetate Ointment, and rinsing with 1% Sodium Bicarbonate (avoiding systemic use during visits)
Behavioral: oral hygiene instruction — Instructions and demonstrations for using manual toothbrushes Instructions and demonstrations for using dental floss or interdental brushes

SUMMARY:
The purpose of this clinical trial is to understand whether the combination of periodontal initial treatment under local anesthesia and glucocorticoids can improve the effectiveness of treatment for erosive oral lichen planus. It will also understand the safety of this treatment regimen.

This study is a single-center, parallel-group, randomized self-controlled trial. The researchers will compare the treatment of periodontal initial therapy combined with glucocorticoid therapy under local anesthesia with traditional glucocorticoid therapy to see if the treatment of periodontal initial therapy combined with glucocorticoid therapy under local anesthesia promotes the healing of erosive oral lichen planus.

Participants will:

One side received periodontal initial treatment combined with glucocorticoid under local anesthesia, while the other side received traditional glucocorticoid therapy Clinical examination at 2, 4, 8, and 12 weeks after treatment Note down the size of their erosion lesion area and periodontal clinical parameters

ELIGIBILITY:
Inclusion Criteria:

* Existence of erosive oral lichen planus that lasts for more than 2 months
* Erosive lesions are located in the buccal mucosa and gingival buccal sulcus of the bilateral mandibular posterior teeth area
* The erosive lesions are mild to moderate (single or multiple small area erosions; 3mm ≤ longest diameter ≤ 10mm; 9mm2 ≤ total area of erosions ≤ 100mm2), and the degree of erosion on both sides is similar (the difference in the size of erosion on both sides does not exceed ± 25%)
* The plaque index in the area of erosive lesions is ≥ 3; Dental calculus index ≥ 2; Gingival index ≥ 2;
* Accompanied by stage II-IV extensive periodontitis

Exclusion Criteria:

* Pregnant women, lactating women, or women planning to conceive during the trial period
* Patients with coagulation dysfunction or other uncontrolled systemic diseases who cannot undergo periodontal treatment
* Has undergone basic periodontal treatment within the past 6 months
* Individuals with a history of allergy to local anesthetic drugs such as articaine
* Individuals with contraindications to glucocorticoids
* Patients with lesion area erosion caused by trauma or chemical stimulation
* Patients with mental disorders who are difficult to cooperate with treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
The erosion area of oral lichen planus | 3 months
  The erosion area of oral lichen planus

SECONDARY OUTCOMES:
visual analogue scale | 2, 4, 8, and 12 weeks
  Mark a horizontal line of 0-10cm on paper with a ruler, and determine the score in millimeters (mm). The score range is 0-100mm, with higher scores indicating greater pain intensity
Clinical score of oral lichen planus | 2, 4, 8, and 12 weeks
probing depth | 4, 8, and 12 weeks
clinical attachment loss | 4, 8, and 12 weeks
plaque index | 4, 8, and 12 weeks
Full mouth bleeding scores | 4, 8, and 12 weeks

OTHER OUTCOMES:
complication | 2, 4, 8, and 12 weeks
  Infection, bleeding, liver and kidney damage, difficulty eating due to pain

CONTACTS AND LOCATIONS:
Overall Officials: Linjun Shi, Doctor, Principal Investigator — Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen H, Shi L, Shang Q, Wei Z, Yang Q, He Y, Li C, Zhou Z, Tang G, Sun H, Awuti G, Song Z, Shi L. Efficacy and safety of periodontal initial therapy combined with intralesional betamethasone sodium phosphate injection under local anesthesia in managing erosive oral lichen planus: study protocol for a multi-center, split-mouth, randomized self-controlled trial. Trials. 2025 Dec 22;26(1):589. doi: 10.1186/s13063-025-09340-5. PMID 41430296